CLINICAL TRIAL: NCT01565642
Title: Goals of Care: A Nursing Home Trial of Decision Support for Advanced Dementia
Acronym: GOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 10-0699; R01AG037483 (NIH)
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Results first posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2016-03

CONDITIONS: Dementia
Keywords: Dementia, decision making
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Decision support intervention (Experimental): Decision aid and care plan meeting
  Interventions: Behavioral: Goals of care decision support
- Control (No Intervention): Attention control information on dementia care

INTERVENTIONS:
Behavioral: Goals of care decision support — Decision aid and care plan meeting
  Arms: Decision support intervention

SUMMARY:
This cluster randomized controlled trial is to examine whether decision support for goals of care can improve quality of communication and decision-making and improve the quality of palliative care for nursing home residents with advanced dementia.

ELIGIBILITY:
Inclusion Criteria:

* Surrogate for nursing home resident with advanced dementia, paired with resident with advanced dementia

Exclusion Criteria:

* Non-related legal surrogate without personal knowledge of resident

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 302 (Actual)
Dates: Start 2012-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura C Hanson, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Ernecoff NC, Zimmerman S, Mitchell SL, Song MK, Lin FC, Wessell KL, Hanson LC. Concordance between Goals of Care and Treatment Decisions for Persons with Dementia. J Palliat Med. 2018 Oct;21(10):1442-1447. doi: 10.1089/jpm.2018.0103. Epub 2018 Jun 29. PMID 29957095
- [Derived] Hanson LC, Zimmerman S, Song MK, Lin FC, Rosemond C, Carey TS, Mitchell SL. Effect of the Goals of Care Intervention for Advanced Dementia: A Randomized Clinical Trial. JAMA Intern Med. 2017 Jan 1;177(1):24-31. doi: 10.1001/jamainternmed.2016.7031. PMID 27893884
- [Derived] Hanson LC, Song MK, Zimmerman S, Gilliam R, Rosemond C, Chisholm L, Lin FC. Fidelity to a behavioral intervention to improve goals of care decisions for nursing home residents with advanced dementia. Clin Trials. 2016 Dec;13(6):599-604. doi: 10.1177/1740774516650863. Epub 2016 Jun 7. PMID 27271683

RESULTS

PARTICIPANT FLOW:
Recruitment Details: April 2012 to September 2014 enrolled dyads of persons with advanced dementia and family decision-makers from 22 participating nursing home sites.
Units Other Than Participants: nursing homes
Period: Overall Study
Arm/Group | Decision Support Intervention | Control
Started | 151; 11 nursing homes | 151; 11 nursing homes
Completed | 149; 11 nursing homes | 150; 11 nursing homes
Not Completed | 2; 0 nursing homes | 1; 0 nursing homes
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Decision Support Intervention | Control | Total
Number analyzed (Participants) | 151 | 151 | 302
Age, Continuous [Mean (Standard Deviation); unit: years] | 85.7 (7.6) | 87.3 (6.7) | 86.5 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 125 | 246
  Male | 30 | 26 | 56
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: African American | 14 | 25 | 39
  Race: White | 134 | 123 | 257
  Race: Other | 3 | 3 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 151 | 151 | 302
Dementia Stage: Global Deterioration Scale (GDS) [Count of Participants; unit: Participants] — The Global deterioration scale includes seven different diagnostic stages ranging between "no cognitive deterioration" and "very serious cognitive deterioration." It investigates the cognitive impairment. Scores range between 1 (no cognitive deterioration) and 7 (very severe cognitive decline) with higher scores reflecting greater severity of cognitive deterioration.
  Participants
    GDS 5 | 38 | 36 | 74
    GDS 6 | 79 | 73 | 152
    GDS 7 | 34 | 42 | 76

OUTCOME MEASURES:

1. Primary Outcome: Quality of Communication and Decision-making
Description: The Quality of Communication (QOC) score with its End of Life (EOL) subscale score. Scores range 0-10 on QOC and its subscales, with higher scores indicating better communication quality.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Decision Support Intervention | Control
Number analyzed (Participants) | 149 | 150
units on a scale
  QOC score | 6.0 (2.0) | 5.6 (1.8)
  QOC End of Life score | 3.7 (2.7) | 3.0 (2.6)

2. Secondary Outcome: Number of Palliative Care Domains in Care Plan
Description: Index score ranging from 0-10 with one point given for care plan addressing each domain: prognosis, goals of care, physical symptoms, emotional needs, spiritual needs, resuscitation, artificial feeding, intravenous fluids, antibiotics, hospitalization. Higher scores indicate better palliative care.
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Decision Support Intervention | Control
Number analyzed (Participants) | 149 | 150
units on a scale | 5.9 (2.2) | 5.3 (1.9)

3. Secondary Outcome: Satisfaction With Care
Description: Satisfaction with Care at the End of Life in Dementia (SWC-EOLD) scale; 10 items rated 1-4 and summed with total potential range 10-40. Higher scores indicate better satisfaction.
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Decision Support Intervention | Control
Number analyzed (Participants) | 149 | 150
units on a scale | 31.0 (5.9) | 31.6 (5.3)

4. Secondary Outcome: Comfort in Dying
Description: Comfort Assessment in Dying for Dementia (CAD-EOLD) includes 14 items rated on a 3 point scale, summed for a total potential score of 14-42. Higher scores indicate better comfort.
Time Frame: 9 months
Population: Decedents only--this outcome measure applies only to residents who die during Follow-Up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Decision Support Intervention | Control
Number analyzed (Participants) | 27 | 33
units on a scale | 34.0 (5.7) | 32.7 (5.4)

5. Secondary Outcome: Alzheimer Disease Related Quality of Life
Description: The Alzheimer Disease Related Quality of Life scale (ADRQL) ranges from 0-100 with higher scores indicating better quality of life.
Time Frame: 9 months
Population: This measure applies only to those persons with dementia who remained alive through the 9 month follow-up. In addition there were 3 withdrawals from the study by 9 months. Thus the overall number of participants for this outcome measure are n=239 (n=302 after removal of 60 decedents and 3 withdrawn participants).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Decision Support Intervention | Control
Number analyzed (Participants) | 122 | 117
units on a scale | 67.8 (15.9) | 65.9 (16.8)

6. Secondary Outcome: Quality of Dying
Description: Quality of Dying in Long-term Care (QOD-LTC) instrument has 11 items in 3 subscales measuring personhood, closure and preparation for dying, for total scores ranging 5-55. Higher scores indicate better quality of the dying experience.
Time Frame: 9 months
Population: Decedents only--this measure applies only to residents who die during Follow-Up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Decision Support Intervention | Control
Number analyzed (Participants) | 27 | 33
units on a scale | 41.7 (7.1) | 41.7 (7.1)

7. Secondary Outcome: Frequency of Communication
Description: Number of participants who report discussions of goals of care with providers -- physicians, nurse practitioners, physician assistants or nursing home staff -- counted during follow-up
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Decision Support Intervention | Control
Number analyzed (Participants) | 149 | 150
Participants | 121 | 123

8. Secondary Outcome: Hospice Referral
Description: Number of participants with a referral to hospice services
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Decision Support Intervention | Control
Number analyzed (Participants) | 149 | 150
Participants | 17 | 18

9. Secondary Outcome: Hospitalizations
Description: Number and timing of transfer to hospital from nursing home care, measured as hospital transfers per 90 person-days of follow-up, with follow-up censored at death.
Time Frame: 9 months
Measure: Number; unit: Hospital transfers per 90 person-days
Arm/Group | Decision Support Intervention | Control
Number analyzed (Participants) | 149 | 150
Hospital transfers per 90 person-days | 0.08 | 0.16

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Decision Support Intervention | Control
All-Cause Mortality (participants affected / at risk) | 27/151 | 33/151
Serious Adverse Events (participants affected / at risk) | 0/151 | 0/151
Other Adverse Events (participants affected / at risk) | 0/151 | 0/151

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No